CLINICAL TRIAL: NCT03316404
Title: Evaluating Multiple Sclerosis Patients ShOWing A GEnomic Signature of Therapy Response
Acronym: EMPOWER
Status: Completed | Type: Observational
Sponsor: DxTerity Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: DXT-MCD-AD02
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis; MS
Keywords: Multiple Sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1 of the study will collect blood samples from participants in various states of the disease. After qualification and informed consent, accepted participants will be sent a blood collection kit and will be asked to complete a study-related questionnaire.
- Cohort 2: Cohort 2 may be conducted at selected clinical sites where MS treatment-naïve patients who are entering a new treatment paradigm will be sought. At the clinical site, patients will be qualified, consented, and a small amount (up to 1mL) of blood will be collected. Between approximately 1 week and 6 months of treatment on the new drug, the participant will be sent another blood collection kit for microsample collection and a brief questionnaire at home. A final sample will be collected between 3 and 6 months after the start of treatment. Within 6 months of initiating treatment, the site will be asked to provide information regarding the health and treatment status of the participant.

SUMMARY:
To develop a test to characterize and monitor Multiple Sclerosis (MS) disease status and therapy response from a participant's home by analyzing the gene expression from participant self-collected blood samples using a novel fingerstick collection kit.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an autoimmune disease that damages the central nervous system (CNS) and disrupts communication to and from the brain by attacking the myelin sheath surrounding neurons. It impairs control of bodily functions and leads to clinical disability as the disease progresses. The worldwide population is estimated at 2.5 million. MS typically develops in young adults; primarily women in their early 30s. The etiology of MS is not fully understood, but it is noted that the prevalence of MS differs with geography and ethnicity.

Biomarker signature panels are important tools for monitoring treatment response and screening for individuals who are unlikely to benefit from certain therapies. To establish a baseline and further characterize gene expression in MS, blood samples from individuals with MS will be collected. A rapid blood test to predict a treatment response would be an innovative diagnostic product that could aid in identifying individuals that may benefit from the targeted therapy. In the long term, such a test could bring significant clinical benefits by enabling individualized treatment to better control the disease, unburdening healthcare costs, and dramatically improving the management of MS.

In order to analyze gene expression data from individuals diagnosed with MS, the study will collect blood samples and information from up to 1500 subjects for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 or older
* Have a permanent address in the United States for the duration of the study
* Have an email address and access to the internet for the duration of the study
* Able to provide informed consent
* Self-reported diagnosis of MS

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with Multiple Sclerosis (MS)
Sampling Method: Non-Probability Sample
Enrollment: 1168 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Obtain blood samples and associated clinical and demographic data from participants diagnosed with Multiple Sclerosis (MS) | 2 years
  Obtain blood samples and associated clinical and demographic data from participants diagnosed with Multiple Sclerosis (MS) to develop a blood test to characterize MS status by analyzing gene expression from blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- DxTerity Diagnostics, Compton, California, United States

IPD SHARING:
Plan to Share IPD: No